CLINICAL TRIAL: NCT01723462
Title: How Often Are Pharmacist Recommendations Followed by Emergency Physicians in Emergency Departments?
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, assistant professor, University of Southern Denmark
Other Study IDs: SLB-ED-02-2012
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Pharmacist Recommendations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical pharmacy has played a role in Emergency Departments (ED). The presence of pharmacists have been shown to reduce medication errors and improve the medication history taken at admission. In Denmark a recent study revealed that clinical pharmacists identified medication problems in 25% of all admission to the ED, of which 47 % were considered to be serious.

However, the pharmacist recommendations are of little value if they are not acknowledged or followed by the physicians.

The aim of the present study was to analyze how often and under which circumstances the physicians made use of pharmaceutical recommendations in an ED with a mixed patient population with special attention to those recommendations, which were of significant or disastrous importance.

ELIGIBILITY:
Inclusion Criteria:

- all acute admissions to emergency department who were treated with one or more drugs

Exclusion Criteria:

- children less than 15 years.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all acute admissions to emergency department
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
number of pharmacist recommendations | up to 48 hours after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Kolding Sygehus, Kolding, Denmark

REFERENCES:
- [Derived] Mogensen CB, Olsen I, Thisted AR. Pharmacist advice is accepted more for medical than for surgical patients in an emergency department. Dan Med J. 2013 Aug;60(8):A4682. PMID 23905567